CLINICAL TRIAL: NCT03438409
Title: Improving Functional Ability in Chronic TBI With Intensive Rehabilitation Robotic Gait Training
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Changes in personnel at Institution.
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, Crystal Massie, Assistant Professor, Indiana University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1703719961
Record Dates: First submitted 2017-08-04; First posted 2018-02-19 (Actual); Last update posted 2018-12-06 (Actual); Status verified 2018-12

CONDITIONS: TBI (Traumatic Brain Injury)
MeSH Terms: conditions — Brain Injuries, Traumatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single Arm Study (Experimental): This study has a single arm with repeated baseline measures. This arm will complete the robotic gait training.
  Interventions: Other: Robotic gait training

INTERVENTIONS:
Other: Robotic gait training — Robotic gait training

SUMMARY:
The purpose of this study is to investigate changes in response to robotic gait training in individuals with a traumatic brain injury.

ELIGIBILITY:
Inclusion Criteria:

* over 18 years of age
* traumatic brain injury at least 6 months prior to study

Exclusion Criteria:

* currently receiving outpatient therapy
* medically unstable
* body weight > 150 kgs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2018-07-30 (Actual); Study Completion 2018-07-30 (Actual)

PRIMARY OUTCOMES:
Change in Functional Gait Outcomes | Change from baseline gait speed to post-test up to 6 weeks following the intervention.
  Gait speed will be assessed using a gait mat.
Change in Endurance | Change from baseline distance covered to post-test up to 6 weeks following the intervention.
  Endurance will be assessed using the 6-minute walk test.

SECONDARY OUTCOMES:
Change in balance | Change from baseline balance to post-test up to 6 weeks following the intervention.
  Balance will be assessed using the Berg Balance Scale.

CONTACTS AND LOCATIONS:
Locations (1):
- Indiana University, Indianapolis, Indiana, United States